CLINICAL TRIAL: NCT00316693
Title: A Phase II Study to Assess the Efficacy, Immunogenicity and Safety of GSK Biologicals' HPV-16/18 L1 VLP AS04 (Cervarix TM) Vaccine Administered Intramuscularly According to a 0, 1, 6 Month Schedule in Healthy Japanese Female Subjects Aged 20 - 25 Years.
Brief Title: Human Papillomavirus (HPV) Vaccine (Cervarix TM) Efficacy, Immunogenicity & Safety Trial in Adult Japanese Women With GSK Biologicals HPV-16/18 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104798
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2009-12-16 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Infections, Papillomavirus
Keywords: HPV Vaccine Efficacy
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of GSK Biologicals HPV-16/18 vaccine (Cervarix™) according to a 0, 1, 6-month schedule.
  Interventions: Biological: HPV-16/18 vaccine (Cervarix™)
- Aimmugen Group (Active Comparator): Subjects received 3 doses of Aimmugen™ (Hepatitis A [HAV] vaccine) according to a 0, 1, 6-month schedule.
  Interventions: Biological: Aimmugen™

INTERVENTIONS:
Biological: HPV-16/18 vaccine (Cervarix™) — Intramuscular injection, 3 doses
  Arms: Cervarix Group
Biological: Aimmugen™ — Intramuscular injection, 3 doses
  Arms: Aimmugen Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Indeed, certain oncogenic types of HPV can infect the cervix (part of the uterus or womb). This infection may go away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. This study will evaluate the efficacy in prevention of persistent HPV-16 or HPV-18 cervical infection lasting at least 6 months, the immunogenicity and safety of GSK Biologicals HPV-16/18 vaccine (Cervarix TM ) over 24 months in Japanese adult women aged 20 - 25 years of age at study start. Approximately 1000 study subjects will either receive the HPV vaccine or a control vaccine (Hepatitis A vaccine) administered intramuscularly according to a 0-1-6 month schedule.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The Protocol Posting has been updated to reflect changes as a consequence of an amendment to the protocol. Sections impacted are Official Title of the study and Intervention name.

ELIGIBILITY:
Inclusion criteria :

* Subjects who the investigator/co-investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A Japanese female subject between, and including, 20 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment.
* Healthy subjects as established by medical history and history-oriented clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects must be of non-childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* Subject must have an intact cervix

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine/control within 30 days preceding the first dose of study vaccine/control, or planned use during the study period.
* Pregnant or breastfeeding women. Women must be at least 3 months post-pregnancy and not breastfeeding to enter the study.
* A women planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period, up to 2 months after the last vaccine dose
* previous administration of components of the investigational vaccine
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Routine vaccines may be allowed up to 8 days before the first dose of study vaccine.
* Previous vaccination against HPV.
* History of vaccination against hepatitis A or a known clinical history of hepatitis A disease
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines
* Hypersensitivity to latex
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of having had colposcopy or has planned a colposcopy to evaluate an abnormal cervical cytology (Pap smear) test.
* Heavy bleeding or heavy vaginal discharge such that a pelvic examination can not be performed
* Acute disease at the time of enrolment.
* Oral temperature >= 37.5°C / axillary temperature > 37.5°C.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1046 (Actual)
Dates: Start 2006-04-26; Primary Completion 2009-02-10 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Japan (2):
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Konno R, Dobbelaere KO, Godeaux OO, Tamura S, Yoshikawa H. Immunogenicity, reactogenicity, and safety of human papillomavirus 16/18 AS04-adjuvanted vaccine in Japanese women: interim analysis of a phase II, double-blind, randomized controlled trial at month 7. Int J Gynecol Cancer. 2009 Jul;19(5):905-11. doi: 10.1111/IGC.0b013e3181a23c0e. PMID 19574783
- [Background] Konno R, Tamura S, Dobbelaere K, Yoshikawa H. Efficacy of human papillomavirus 16/18 AS04-adjuvanted vaccine in Japanese women aged 20 to 25 years: interim analysis of a phase 2 double-blind, randomized, controlled trial. Int J Gynecol Cancer. 2010 Apr;20(3):404-10. doi: 10.1111/IGC.0b013e3181d373a5. PMID 20375805
- [Background] Konno R, Tamura S, Dobbelaere K, Yoshikawa H. Prevalence and type distribution of human papillomavirus in healthy Japanese women aged 20 to 25 years old enrolled in a clinical study. Cancer Sci. 2011 Apr;102(4):877-82. doi: 10.1111/j.1349-7006.2011.01878.x. Epub 2011 Feb 17. PMID 21251162
- [Background] Konno R et al. Efficacy, immunogenicity and safety of HPV 16/18 AS04-adjuvanted vaccine in Japanese women. Abstract presented at European Research Organization on Genital Infection and Neoplasia 2010 (EUROGIN). Monte Carlo, Monaco, 17-20 February 2010.
- [Background] Konno R et al. Interim analysis of clinical trial of HPV-16/18-AS04 vaccine in Japan. Abstract presented at the 25th International Papillomavirus Conference, Malmö, Sweden, 8-14 May 2009.
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Chen J, Gopala K, Akarsh PK, Struyf F, Rosillon D. Prevalence and Incidence of Human Papillomavirus (HPV) Infection Before and After Pregnancy: Pooled Analysis of the Control Arms of Efficacy Trials of HPV-16/18 AS04-Adjuvanted Vaccine. Open Forum Infect Dis. 2019 Dec 4;6(12):ofz486. doi: 10.1093/ofid/ofz486. eCollection 2019 Dec. PMID 31824976
- [Derived] Konno R, Yoshikawa H, Okutani M, Quint W, V Suryakiran P, Lin L, Struyf F. Efficacy of the human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical intraepithelial neoplasia and cervical infection in young Japanese women. Hum Vaccin Immunother. 2014;10(7):1781-94. doi: 10.4161/hv.28712. PMID 25424783
- [Derived] Konno R, Tamura S, Dobbelaere K, Yoshikawa H. Efficacy of human papillomavirus type 16/18 AS04-adjuvanted vaccine in Japanese women aged 20 to 25 years: final analysis of a phase 2 double-blind, randomized controlled trial. Int J Gynecol Cancer. 2010 Jul;20(5):847-55. doi: 10.1111/IGC.0b013e3181da2128. PMID 20606533
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six subjects enrolled in this study were not vaccinated and hence not reported as started in the participant flow table below.
Period: Overall Study
Arm/Group | Cervarix Group | Aimmugen Group
Started | 519 | 521
Completed | 442 | 436
Not Completed | 77 | 85
Not completed — Adverse Event | 6 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 26 | 34
Not completed — Other | 38 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Aimmugen Group | Total
Number analyzed (Participants) | 519 | 521 | 1040
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (1.7) | 22.5 (1.6) | 22.5 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519 | 521 | 1040
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese heritage | 519 | 521 | 1040

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Persistent Cervical Infection With Human Papillomavirus 16 (HPV-16) or Human Papillomavirus 18 (HPV-18)
Description: Persistent HPV-16 or HPV-18 infection is defined as at least 2 positive Human Papillomavirus (HPV) deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assays for the same viral genotype with no negative DNA sample between the 2 positive DNA samples, over an approximate interval of 6 months (> 150 days) [as assessed in women who were, for the corresponding HPV type, seronegative at Month 0 and HPV DNA negative (by PCR) at Month 0 and Month 6].
Time Frame: Throughout the study period (up to Month 24)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 387 | 392
Participants
  HPV-16/18 | 0 | 15
  HPV-16: number analyzed (Participants) | 332 | 340
  HPV-16 | 0 | 11
  HPV-18: number analyzed (Participants) | 346 | 343
  HPV-18 | 0 | 5

2. Secondary Outcome: Number of Subjects With Incident Cervical Infection With Human Papillomavirus 16 (HPV-16) or Human Papillomavirus 18 (HPV-18)
Description: HPV-16 or HPV-18 incident infection is defined as at least one positive HPV-16 or HPV-18 deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assay in women who were, for the corresponding HPV type, seronegative at Month 0 and HPV DNA negative (by PCR) at Month 0 and Month 6.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 408 | 406
Participants
  HPV-16/18 | 7 | 39
  HPV-16: number analyzed (Participants) | 351 | 353
  HPV-16 | 4 | 22
  HPV-18: number analyzed (Participants) | 359 | 355
  HPV-18 | 3 | 18

3. Secondary Outcome: Number of Subjects With Cytologically-confirmed Abnormalities Concurrently Associated With Human Papillomavirus 16 (HPV-16) and/or Human Papillomavirus 18 (HPV-18) Cervical Infection
Description: Cytologically-confirmed abnormalities assessed include atypical squamous cells of undetermined significance (ASC-US), low-grade squamous intraepithelial lesion (LSIL), high-grade squamous intraepithelial lesion (HSIL), atypical squamous cells-can not exclude HSIL (ASC-H) and atypical glandular cells (AGC). These cytological abnormalities were assessed in women who were, for the corresponding Human Papillomavirus (HPV) type, seronegative at Month 0 and HPV deoxyribonucleic acid (DNA) negative (by polymerase chain reaction) at Month 0 and Month 6.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 408 | 406
Participants
  HPV-16/18 | 1 | 12
  HPV-16: number analyzed (Participants) | 351 | 353
  HPV-16 | 0 | 8
  HPV-18: number analyzed (Participants) | 359 | 355
  HPV-18 | 1 | 4

4. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Lesions Concurrently Associated With Human Papillomavirus 16 (HPV-16) and/or Human Papillomavirus (HPV-18) Cervical Infection
Description: Histopathologically-confirmed lesions assessed include cervical intraepithelial neoplasia of grade 1 (CIN1), grade 2 (CIN2), grade 3 (CIN3) and adenocarcinoma. These lesions were assessed in women who were, for the corresponding Human Papillomavirus (HPV) type, seronegative at Month 0 and HPV deoxyribonucleic acid (DNA) negative (by polymerase chain reaction) at Month 0 and Month 6.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 408 | 407
Participants
  HPV-16/18 | 0 | 3
  HPV-16: number analyzed (Participants) | 351 | 353
  HPV-16 | 0 | 2
  HPV-18: number analyzed (Participants) | 359 | 356
  HPV-18 | 0 | 1

5. Secondary Outcome: Number of Subjects With Incident Cervical Infection With Any Oncogenic Human Papillomavirus (HPV) Types
Description: Incident infection for oncogenic HPV types is defined as at least one positive oncogenic HPV type deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assay in women who were, for the corresponding HPV type, HPV DNA negative (by PCR) at Month 0 and Month 6.
  Oncogenic (high risk [HR]) HPV types assessed include HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 446 | 436
Participants
  HPV-16: number analyzed (Participants) | 119 | 398
  HPV-16 | 5 | 24
  HPV-18: number analyzed (Participants) | 428 | 407
  HPV-18 | 4 | 20
  HPV-31: number analyzed (Participants) | 428 | 416
  HPV-31 | 8 | 7
  HPV-33: number analyzed (Participants) | 444 | 435
  HPV-33 | 2 | 5
  HPV-35: number analyzed (Participants) | 443 | 432
  HPV-35 | 7 | 4
  HPV-39: number analyzed (Participants) | 422 | 418
  HPV-39 | 13 | 14
  HPV-45: number analyzed (Participants) | 446 | 433
  HPV-45 | 0 | 0
  HPV-51: number analyzed (Participants) | 413 | 412
  HPV-51 | 14 | 29
  HPV-52: number analyzed (Participants) | 404 | 383
  HPV-52 | 30 | 32
  HPV-56: number analyzed (Participants) | 423 | 414
  HPV-56 | 15 | 15
  HPV-58: number analyzed (Participants) | 432 | 411
  HPV-58 | 12 | 13
  HPV-59: number analyzed (Participants) | 443 | 427
  HPV-59 | 8 | 5
  HPV-66: number analyzed (Participants) | 426 | 410
  HPV-66 | 6 | 13
  HPV-68: number analyzed (Participants) | 436 | 424
  HPV-68 | 8 | 12
  Any HR HPV types except HPV-16/18 | 90 | 113
  Any HR HPV types | 98 | 134

6. Secondary Outcome: Number of Subjects With Persistent Cervical Infection With Any Oncogenic Human Papillomavirus (HPV) Types
Description: Persistent infection for oncogenic HPV types is defined as at least 2 positive HPV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assays for the same viral genotype with no negative DNA sample between the 2 positive DNA samples, over an approximate interval of 6 months (> 150 days) [as assessed in women who were, for the corresponding HPV type, HPV DNA negative (by PCR) at Month 0 and Month 6].
  Oncogenic (high risk [HR]) HPV types assessed include HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 424 | 422
Participants
  HPV-16: number analyzed (Participants) | 398 | 384
  HPV-16 | 0 | 12
  HPV-18: number analyzed (Participants) | 408 | 394
  HPV-18 | 0 | 5
  HPV-31: number analyzed (Participants) | 406 | 403
  HPV-31 | 4 | 2
  HPV-33: number analyzed (Participants) | 422 | 421
  HPV-33 | 0 | 2
  HPV-35: number analyzed (Participants) | 422 | 418
  HPV-35 | 1 | 1
  HPV-39: number analyzed (Participants) | 401 | 406
  HPV-39 | 2 | 4
  HPV-45: number analyzed (Participants) | 424 | 419
  HPV-45 | 0 | 0
  HPV-51: number analyzed (Participants) | 395 | 398
  HPV-51 | 5 | 10
  HPV-52: number analyzed (Participants) | 393 | 371
  HPV-52 | 11 | 5
  HPV-56: number analyzed (Participants) | 403 | 400
  HPV-56 | 4 | 7
  HPV-58: number analyzed (Participants) | 410 | 399
  HPV-58 | 4 | 8
  HPV-59: number analyzed (Participants) | 422 | 413
  HPV-59 | 1 | 0
  HPV-66: number analyzed (Participants) | 404 | 396
  HPV-66 | 0 | 3
  HPV-68: number analyzed (Participants) | 415 | 410
  HPV-68 | 2 | 1
  Any HR HPV types except HPV-16/18 | 27 | 39
  Any HR HPV types | 27 | 53

7. Secondary Outcome: Number of Subjects With Cytologically-confirmed Abnormalities Concurrently Associated With Cervical Infection With Any Oncogenic Human Papillomavirus (HPV) Type
Description: Cytologically-confirmed abnormalities assessed include ASC-US, LSIL, HSIL, ASC-H and AGC. These cytological abnormalities were assessed in women who were, for the corresponding HPV type (determined by PCR), HPV DNA negative (by PCR) at Month 0 and Month 6.
  Oncogenic (high risk [HR]) HPV types assessed include HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 446 | 436
Participants
  HPV-16: number analyzed (Participants) | 419 | 398
  HPV-16 | 0 | 9
  HPV-18: number analyzed (Participants) | 428 | 407
  HPV-18 | 1 | 4
  HPV-31: number analyzed (Participants) | 428 | 416
  HPV-31 | 2 | 0
  HPV-33: number analyzed (Participants) | 444 | 435
  HPV-33 | 1 | 2
  HPV-35: number analyzed (Participants) | 443 | 432
  HPV-35 | 2 | 1
  HPV-39: number analyzed (Participants) | 422 | 418
  HPV-39 | 3 | 5
  HPV-45: number analyzed (Participants) | 446 | 433
  HPV-45 | 0 | 0
  HPV-51: number analyzed (Participants) | 413 | 412
  HPV-51 | 4 | 5
  HPV-52: number analyzed (Participants) | 404 | 383
  HPV-52 | 6 | 7
  HPV-56: number analyzed (Participants) | 423 | 414
  HPV-56 | 5 | 6
  HPV-58: number analyzed (Participants) | 432 | 411
  HPV-58 | 4 | 10
  HPV-59: number analyzed (Participants) | 443 | 427
  HPV-59 | 3 | 3
  HPV-66: number analyzed (Participants) | 426 | 410
  HPV-66 | 1 | 3
  HPV-68: number analyzed (Participants) | 436 | 424
  HPV-68 | 3 | 5
  Any HR HPV types except HPV-16/18 | 23 | 35
  Any HR HPV types | 24 | 42

8. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Lesions Concurrently Associated With Cervical Infection With Any Oncogenic Human Papillomavirus (HPV) Type
Description: Histopathologically-confirmed lesions assessed include cervical intraepithelial neoplasia of grade 1 (CIN1), grade 2 (CIN2), grade 3 (CIN3) and adenocarcinoma. These lesions were assessed in women who were, for the corresponding HPV type (determined by polymerase chain reaction)), HPV deoxyribonucleic acid (DNA) negative at Month 0 and Month 6.
  Oncogenic (high risk [HR]) HPV types assessed include HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68.
Time Frame: Up to Month 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 446 | 438
Participants
  HPV-16: number analyzed (Participants) | 419 | 400
  HPV-16 | 0 | 3
  HPV-18: number analyzed (Participants) | 428 | 409
  HPV-18 | 0 | 1
  HPV-31: number analyzed (Participants) | 428 | 417
  HPV-31 | 0 | 0
  HPV-33: number analyzed (Participants) | 444 | 437
  HPV-33 | 0 | 1
  HPV-35: number analyzed (Participants) | 443 | 434
  HPV-35 | 0 | 0
  HPV-39: number analyzed (Participants) | 422 | 419
  HPV-39 | 0 | 1
  HPV-45: number analyzed (Participants) | 446 | 435
  HPV-45 | 0 | 0
  HPV-51: number analyzed (Participants) | 413 | 413
  HPV-51 | 2 | 2
  HPV-52: number analyzed (Participants) | 404 | 385
  HPV-52 | 3 | 5
  HPV-56: number analyzed (Participants) | 423 | 415
  HPV-56 | 0 | 0
  HPV-58: number analyzed (Participants) | 432 | 413
  HPV-58 | 1 | 5
  HPV-59: number analyzed (Participants) | 443 | 429
  HPV-59 | 0 | 1
  HPV-66: number analyzed (Participants) | 426 | 412
  HPV-66 | 0 | 0
  HPV-68: number analyzed (Participants) | 436 | 425
  HPV-68 | 0 | 2
  Any HR HPV types except HPV-16/18 | 6 | 14
  Any HR HPV types | 6 | 17

9. Secondary Outcome: Number of Subjects With Anti-human Papillomavirus 16 and 18 (Anti-HPV-16 and Anti-HPV-18) Antibody Titers Above the Cut-off Value
Description: Anti-HPV-16 antibody cut-off value assessed include 8 ELISA units per milliliter (EL.U/mL) and anti-HPV-18 antibody cut-off value assessed include 7 EL.U/mL.
Time Frame: At Months 0 (pre-vaccination), 6, 7, 12, 18 and 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 411 | 393
Participants
  HPV-16 (pre-vaccination) | 64 | 51
  HPV-16 (Month 6) | 411 | 55
  HPV-16 (Month 7): number analyzed (Participants) | 410 | 387
  HPV-16 (Month 7) | 410 | 52
  HPV-16 (Month 12): number analyzed (Participants) | 373 | 334
  HPV-16 (Month 12) | 373 | 46
  HPV-16 (Month 18): number analyzed (Participants) | 356 | 307
  HPV-16 (Month 18) | 356 | 39
  HPV-16 (Month 24): number analyzed (Participants) | 351 | 295
  HPV-16 (Month 24) | 351 | 38
  HPV-18 (pre-vaccination): number analyzed (Participants) | 410 | 390
  HPV-18 (pre-vaccination) | 61 | 48
  HPV-18 (Month 6): number analyzed (Participants) | 410 | 388
  HPV-18 (Month 6) | 410 | 53
  HPV-18 (Month 7): number analyzed (Participants) | 409 | 385
  HPV-18 (Month 7) | 409 | 54
  HPV-18 (Month 12): number analyzed (Participants) | 372 | 329
  HPV-18 (Month 12) | 372 | 55
  HPV-18 (Month 18): number analyzed (Participants) | 355 | 302
  HPV-18 (Month 18) | 355 | 40
  HPV-18 (Month 24): number analyzed (Participants) | 350 | 288
  HPV-18 (Month 24) | 350 | 38

10. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Months 0, 6, 7, 12, 18 and 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 411 | 393
EL.U/mL
  Anti-HPV-16 (Month 0) | 5.5 [5.1 to 5.9] | 5.3 [4.9 to 5.7]
  Anti-HPV-16 (Month 6) | 708.4 [650.1 to 772.0] | 5.4 [4.9 to 5.8]
  Anti-HPV-16 (Month 7): number analyzed (Participants) | 410 | 387
  Anti-HPV-16 (Month 7) | 7441.0 [6854.3 to 8077.8] | 5.3 [4.9 to 5.8]
  Anti-HPV-16 (Month 12): number analyzed (Participants) | 373 | 334
  Anti-HPV-16 (Month 12) | 2877.7 [2623.1 to 3156.9] | 5.3 [4.9 to 5.8]
  Anti-HPV-16 (Month 18): number analyzed (Participants) | 356 | 307
  Anti-HPV-16 (Month 18) | 1864.8 [1694.5 to 2052.2] | 5.3 [4.8 to 5.8]
  Anti-HPV-16 (Month 24): number analyzed (Participants) | 351 | 295
  Anti-HPV-16 (Month 24) | 1532.2 [1395.1 to 1682.7] | 5.4 [4.9 to 5.9]
  Anti-HPV-18 (Month 0): number analyzed (Participants) | 410 | 390
  Anti-HPV-18 (Month 0) | 4.5 [4.2 to 4.8] | 4.4 [4.1 to 4.7]
  Anti-HPV-18 (Month 6): number analyzed (Participants) | 410 | 388
  Anti-HPV-18 (Month 6) | 504.6 [464.6 to 548.1] | 4.4 [4.1 to 4.7]
  Anti-HPV-18 (Month 7): number analyzed (Participants) | 409 | 385
  Anti-HPV-18 (Month 7) | 3805.4 [3515.6 to 4119.1] | 4.5 [4.2 to 4.8]
  Anti-HPV-18 (Month 12): number analyzed (Participants) | 372 | 329
  Anti-HPV-18 (Month 12) | 1330.7 [1210.2 to 1463.2] | 4.5 [4.2 to 4.8]
  Anti-HPV-18 (Month 18): number analyzed (Participants) | 355 | 302
  Anti-HPV-18 (Month 18) | 782.0 [703.4 to 869.5] | 4.4 [4.1 to 4.7]
  Anti-HPV-18 (Month 24): number analyzed (Participants) | 350 | 288
  Anti-HPV-18 (Month 24) | 627.8 [566.3 to 696.0] | 4.4 [4.1 to 4.8]

11. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include arthralgia, fatigue, fever (above 37.5 degree Celsius), gastrointestinal symptoms, headache, myalgia, rash and urticaria.
Time Frame: Within 7 days after each and any vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 512 | 511
Participants
  Pain: number analyzed (Participants) | 512 | 510
  Pain | 508 | 214
  Redness: number analyzed (Participants) | 512 | 510
  Redness | 455 | 287
  Swelling: number analyzed (Participants) | 512 | 510
  Swelling | 401 | 165
  Arthralgia | 123 | 61
  Fatigue | 341 | 300
  Fever | 41 | 28
  Gastro-intestinal symptoms | 172 | 167
  Headache | 250 | 222
  Myalgia | 262 | 128
  Rash | 33 | 24
  Urticaria | 16 | 20

12. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 30 days after any vaccination
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants | 294 | 266

13. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (up to Month 24)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants | 18 | 19

14. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Other Medically Significant Conditions (MSCs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. MSC include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Throughout the study period (up to Month 24)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants
  NOCDs | 5 | 6
  MSCs | 91 | 107

15. Secondary Outcome: Outcome of Any Reported Pregnancies
Description: Information on any subject who became pregnant while participating in this study was collected. The outcomes of the pregnancies are reported below.
Time Frame: Throughout the study period (up to Month 24)
Population: Analysis was performed on those subjects reporting pregnancy during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 46 | 43
Participants
  Normal infant | 20 | 19
  Premature birth | 1 | 0
  Elective termination | 14 | 16
  Spontaneous abortion | 5 | 3
  Lost to follow-up | 1 | 0
  Pregnancy ongoing | 5 | 5

16. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Hematological Parameters
Description: Hematological parameters assessed in blood samples include hemoglobin, haematocrit, mean corpuscular (MC) hemoglobin, mean corpuscular (MC) hemoglobin concentration, mean corpuscular (MC) volume, platelet count, red blood cell count, white blood cell count.
  Abnormalities reported include values outside the normal ranges: values higher than normal are designated as "Above" and values lower than normal as "Below" while "Unknown" stands for values not determined.
Time Frame: At Month 0 and Month 7
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants
  Hemoglobin Normal [Month 0] | 499 | 498
  Hemoglobin Above [Month 0] | 1 | 2
  Hemoglobin Below [Month 0] | 18 | 21
  Hemoglobin Unknown [Month 0] | 1 | 0
  Hemoglobin Normal [Month 7] | 448 | 444
  Hemoglobin Above [Month 7] | 7 | 7
  Hemoglobin Below [Month 7] | 12 | 22
  Hemoglobin Unknown [Month 7] | 52 | 48
  Hematocrit Normal [Month 0] | 501 | 506
  Hematocrit Above [Month 0] | 3 | 5
  Hematocrit Below [Month 0] | 14 | 10
  Hematocrit Unknown [Month 0] | 1 | 0
  Hematocrit Normal [Month 7] | 448 | 456
  Hematocrit Above [Month 7] | 11 | 4
  Hematocrit Below [Month 7] | 8 | 13
  Hematocrit Unknown [Month 7] | 52 | 48
  Platelet count Normal [Month 0] | 504 | 514
  Platelet count Above [Month 0] | 13 | 5
  Platelet count Below [Month 0] | 0 | 2
  Platelet count Unknown [Month 0] | 2 | 0
  Platelet count Normal [Month 7] | 456 | 461
  Platelet count Above [Month 7] | 9 | 10
  Platelet count Below [Month 7] | 1 | 2
  Platelet count Unknown [Month 7] | 53 | 48
  Red Blood Cells count Normal [Month 0] | 514 | 515
  Red Blood Cells count Above [Month 0] | 2 | 4
  Red Blood Cells count Below [Month 0] | 2 | 2
  Red Blood Cells count Unknown [Month 0] | 1 | 0
  Red Blood Cells count Normal [Month 7] | 457 | 463
  Red Blood Cells count Above [Month 7] | 6 | 5
  Red Blood Cells count Below [Month 7] | 4 | 5
  Red Blood Cells count Unknown [Month 7] | 52 | 48
  White Blood Cells count Normal [Month 0] | 496 | 499
  White Blood Cells count Above [Month 0] | 12 | 14
  White Blood Cells count Below [Month 0] | 10 | 8
  White Blood Cells count Unknown [Month 0] | 1 | 0
  White Blood Cells count Normal [Month 7] | 440 | 453
  White Blood Cells count Above [Month 7] | 23 | 16
  White Blood Cells count Below [Month 7] | 4 | 4
  White Blood Cells count Unknown [Month 7] | 52 | 48
  MC hemoglobin Normal [Month 0] | 489 | 491
  MC hemoglobin Above [Month 0] | 0 | 0
  MC hemoglobin Below [Month 0] | 29 | 30
  MC hemoglobin Unknown [Month 0] | 1 | 0
  MC hemoglobin Normal [Month 7] | 441 | 439
  MC hemoglobin Above [Month 7] | 0 | 0
  MC hemoglobin Below [Month 7] | 26 | 34
  MC hemoglobin Unknown [Month 7] | 52 | 48
  MC hemoglobin concentration Normal [Month 0] | 495 | 488
  MC hemoglobin concentration Above [Month 0] | 0 | 0
  MC hemoglobin concentration Below [Month 0] | 23 | 33
  MC hemoglobin concentration Unknown [Month 0] | 1 | 0
  MC hemoglobin concentration Normal [Month 7] | 442 | 434
  MC hemoglobin concentration Above [Month 7] | 0 | 0
  MC hemoglobin concentration Below [Month 7] | 25 | 39
  MC hemoglobin concentration Unknown [Month 7] | 52 | 48
  MC volume Normal [Month 0] | 504 | 505
  MC volume Above [Month 0] | 1 | 0
  MC volume Below [Month 0] | 13 | 16
  MC volume Unknown [Month 0] | 1 | 0
  MC volume Normal [Month 7] | 457 | 456
  MC volume Above [Month 7] | 2 | 1
  MC volume Below [Month 7] | 8 | 16
  MC volume Unknown [Month 7] | 52 | 48

17. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical Parameters
Description: Biochemical parameters were assessed in blood samples. Abnormalities reported include values outside the normal ranges: values higher than normal are designated as "Above" and values lower than normal as "Below" while "Unknown" stands for values not determined.
  Abbreviations: aminotransferase (ALT), aspartate aminotransferase (ASP), C reactive protein (CRP), gamma-glutamyl-transferase (GGT) and lactate dehydrogenase (LDH).
Time Frame: At Month 0 and Month 7
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants
  Albumin Normal [Month 0] | 519 | 521
  Albumin Above [Month 0] | 0 | 0
  Albumin Below [Month 0] | 0 | 0
  Albumin Unknown [Month 0] | 0 | 0
  Albumin Normal [Month 7] | 466 | 472
  Albumin Above [Month 7] | 0 | 0
  Albumin Below [Month 7] | 1 | 2
  Albumin Unknown [Month 7] | 52 | 47
  Albumin/Globulin ratio Normal [Month 0] | 483 | 488
  Albumin/Globulin ratio Above [Month 0] | 20 | 20
  Albumin/Globulin ratio Below [Month 0] | 16 | 13
  Albumin/Globulin ratio Unknown [Month 0] | 0 | 0
  Albumin/Globulin ratio Normal [Month 7] | 421 | 443
  Albumin/Globulin ratio Above [Month 7] | 30 | 19
  Albumin/Globulin ratio Below [Month 7] | 16 | 12
  Albumin/Globulin ratio Unknown [Month 7] | 52 | 47
  Alkaline phosphatase Normal [Month 0] | 500 | 497
  Alkaline phosphatase Above [Month 0] | 3 | 4
  Alkaline phosphatase Below [Month 0] | 16 | 20
  Alkaline phosphatase Unknown [Month 0] | 0 | 0
  Alkaline phosphatase Normal [Month 7] | 451 | 453
  Alkaline phosphatase Above [Month 7] | 4 | 3
  Alkaline phosphatase Below [Month 7] | 12 | 18
  Alkaline phosphatase Unknown [Month 7] | 52 | 47
  ALT Normal [Month 0] | 510 | 518
  ALT Above [Month 0] | 8 | 3
  ALT Below [Month 0] | 1 | 0
  ALT Unknown [Month 0] | 0 | 0
  ALT Normal [Month 7] | 457 | 471
  ALT Above [Month 7] | 9 | 3
  ALT Below [Month 7] | 1 | 0
  ALT Unknown [Month 7] | 52 | 47
  AST Normal [Month 0] | 516 | 520
  AST Above [Month 0] | 3 | 1
  AST Below [Month 0] | 0 | 0
  AST Unknown [Month 0] | 0 | 0
  AST Normal [Month 7] | 464 | 472
  AST Above [Month 7] | 3 | 0
  AST Below [Month 7] | 0 | 2
  AST Unknown [Month 7] | 52 | 47
  Blood Urea Nitrogen Normal [Month 0] | 450 | 466
  Blood Urea Nitrogen Above [Month 0] | 7 | 3
  Blood Urea Nitrogen Below [Month 0] | 62 | 52
  Blood Urea Nitrogen Unknown [Month 0] | 0 | 0
  Blood Urea Nitrogen Normal [Month 7] | 417 | 434
  Blood Urea Nitrogen Above [Month 7] | 3 | 1
  Blood Urea Nitrogen Below [Month 7] | 47 | 39
  Blood Urea Nitrogen Unknown [Month 7] | 52 | 47
  Calcium Normal [Month 0] | 516 | 519
  Calcium Above [Month 0] | 3 | 2
  Calcium Below [Month 0] | 0 | 0
  Calcium Unknown [Month 0] | 0 | 0
  Calcium Normal [Month 7] | 461 | 468
  Calcium Above [Month 7] | 3 | 4
  Calcium Below [Month 7] | 3 | 2
  Calcium Unknown [Month 7] | 52 | 47
  Total cholesterol Normal [Month 0] | 407 | 402
  Total cholesterol Above [Month 0] | 42 | 34
  Total cholesterol Below [Month 0] | 70 | 85
  Total cholesterol Unknown [Month 0] | 0 | 0
  Total cholesterol Normal [Month 7] | 355 | 367
  Total cholesterol Above [Month 7] | 36 | 36
  Total cholesterol Below [Month 7] | 76 | 71
  Total cholesterol Unknown [Month 7] | 52 | 47
  Chlorine Normal [Month 0] | 518 | 518
  Chlorine Above [Month 0] | 0 | 1
  Chlorine Below [Month 0] | 1 | 2
  Chlorine Unknown [Month 0] | 0 | 0
  Chlorine Normal [Month 7] | 466 | 472
  Chlorine Above [Month 7] | 0 | 0
  Chlorine Below [Month 7] | 1 | 2
  Chlorine Unknown [Month 7] | 52 | 47
  Creatinine phosphokinase Normal [Month 0] | 456 | 454
  Creatinine phosphokinase Above [Month 0] | 13 | 13
  Creatinine phosphokinase Below [Month 0] | 50 | 54
  Creatinine phosphokinase Unknown [Month 0] | 0 | 0
  Creatinine phosphokinase Normal [Month 7] | 412 | 420
  Creatinine phosphokinase Above [Month 7] | 10 | 7
  Creatinine phosphokinase Below [Month 7] | 45 | 47
  Creatinine phosphokinase Unknown [Month 7] | 52 | 47
  Creatinine Normal [Month 0] | 510 | 509
  Creatinine Above [Month 0] | 2 | 4
  Creatinine Below [Month 0] | 7 | 8
  Creatinine Unknown [Month 0] | 0 | 0
  Creatinine Normal [Month 7] | 453 | 466
  Creatinine Above [Month 7] | 3 | 2
  Creatinine Below [Month 7] | 11 | 6
  Creatinine Unknown [Month 7] | 52 | 47
  Direct bilirubin Normal [Month 0] | 500 | 494
  Direct bilirubin Above [Month 0] | 19 | 27
  Direct bilirubin Below [Month 0] | 0 | 0
  Direct bilirubin Unknown [Month 0] | 0 | 0
  Direct bilirubin Normal [Month 7] | 457 | 458
  Direct bilirubin Above [Month 7] | 10 | 16
  Direct bilirubin Below [Month 7] | 0 | 0
  Direct bilirubin Unknown [Month 7] | 52 | 47
  GGT Normal [Month 0] | 510 | 515
  GGT Above [Month 0] | 9 | 6
  GGT Below [Month 0] | 0 | 0
  GGT Unknown [Month 0] | 0 | 0
  GGT Normal [Month 7] | 459 | 471
  GGT Above [Month 7] | 8 | 3
  GGT Below [Month 7] | 0 | 0
  GGT Unknown [Month 7] | 52 | 47
  Glucose Normal [Month 0] | 468 | 464
  Glucose Above [Month 0] | 10 | 11
  Glucose Below [Month 0] | 41 | 47
  Glucose Unknown [Month 0] | 0 | 0
  Glucose Normal [Month 7] | 409 | 423
  Glucose Above [Month 7] | 15 | 18
  Glucose Below [Month 7] | 43 | 34
  Glucose Unknown [Month 7] | 52 | 47
  Potassium Normal [Month 0] | 509 | 509
  Potassium Above [Month 0] | 10 | 11
  Potassium Below [Month 0] | 0 | 1
  Potassium Unknown [Month 0] | 0 | 0
  Potassium Normal [Month 7] | 462 | 470
  Potassium Above [Month 7] | 5 | 4
  Potassium Below [Month 7] | 0 | 0
  Potassium Unknown [Month 7] | 52 | 47
  Leucine Amino Peptidase Normal [Month 0] | 510 | 512
  Leucine Amino Peptidase Above [Month 0] | 4 | 1
  Leucine Amino Peptidase Below [Month 0] | 5 | 8
  Leucine Amino Peptidase Unknown [Month 0] | 0 | 0
  Leucine Amino Peptidase Normal [Month 7] | 460 | 462
  Leucine Amino Peptidase Above [Month 7] | 2 | 9
  Leucine Amino Peptidase Below [Month 7] | 5 | 3
  Leucine Amino Peptidase Unknown [Month 7] | 52 | 47
  LDH Normal [Month 0] | 486 | 491
  LDH Above [Month 0] | 2 | 1
  LDH Below [Month 0] | 31 | 29
  LDH Unknown [Month 0] | 0 | 0
  LDH Normal [Month 7] | 433 | 437
  LDH Above [Month 7] | 5 | 2
  LDH Below [Month 7] | 29 | 35
  LDH Unknown [Month 7] | 52 | 47
  Sodium Normal [Month 0] | 519 | 521
  Sodium Above [Month 0] | 0 | 0
  Sodium Below [Month 0] | 0 | 0
  Sodium Unknown [Month 0] | 0 | 0
  Sodium Normal [Month 7] | 466 | 474
  Sodium Above [Month 7] | 1 | 0
  Sodium Below [Month 7] | 0 | 0
  Sodium Unknown [Month 7] | 52 | 47
  Total bilirubin Normal [Month 0] | 472 | 466
  Total bilirubin Above [Month 0] | 47 | 55
  Total bilirubin Below [Month 0] | 0 | 0
  Total bilirubin Unknown [Month 0] | 0 | 0
  Total bilirubin Normal [Month 7] | 440 | 443
  Total bilirubin Above [Month 7] | 27 | 31
  Total bilirubin Below [Month 7] | 0 | 0
  Total bilirubin Unknown [Month 7] | 52 | 47
  Triglycerides Normal [Month 0] | 318 | 324
  Triglycerides Above [Month 0] | 24 | 21
  Triglycerides Below [Month 0] | 177 | 176
  Triglycerides Unknown [Month 0] | 0 | 0
  Triglycerides Normal [Month 7] | 275 | 290
  Triglycerides Above [Month 7] | 28 | 26
  Triglycerides Below [Month 7] | 164 | 158
  Triglycerides Unknown [Month 7] | 52 | 47
  Total protein Normal [Month 0] | 510 | 509
  Total protein Above [Month 0] | 6 | 10
  Total protein Below [Month 0] | 3 | 2
  Total protein Unknown [Month 0] | 0 | 0
  Total protein Normal [Month 7] | 454 | 463
  Total protein Above [Month 7] | 1 | 2
  Total protein Below [Month 7] | 12 | 9
  Total protein Unknown [Month 7] | 52 | 47
  Uric acid Normal [Month 0] | 515 | 520
  Uric acid Above [Month 0] | 4 | 1
  Uric acid Below [Month 0] | 0 | 0
  Uric acid Unknown [Month 0] | 0 | 0
  Uric acid Normal [Month 7] | 465 | 473
  Uric acid Above [Month 7] | 2 | 1
  Uric acid Below [Month 7] | 0 | 0
  Uric acid Unknown [Month 7] | 52 | 47
  pH Normal [Month 0] | 466 | 462
  pH Above [Month 0] | 52 | 59
  pH Below [Month 0] | 0 | 0
  pH Unknown [Month 0] | 1 | 0
  pH Normal [Month 7] | 438 | 442
  pH Above [Month 7] | 28 | 32
  pH Below [Month 7] | 0 | 0
  pH Unknown [Month 7] | 53 | 47
  CRP Normal [Month 0] | 106 | 70
  CRP Above [Month 0] | 12 | 11
  CRP Below [Month 0] | 0 | 0
  CRP Unknown [Month 0] | 401 | 440
  CRP Normal [Month 7] | 126 | 96
  CRP Above [Month 7] | 20 | 16
  CRP Below [Month 7] | 0 | 0
  CRP Unknown [Month 7] | 373 | 409

18. Secondary Outcome: Number of Subjects Reporting Abnormal Biochemical Parameters in Urine Samples
Description: Abnormalities in concentrations (expressed as milligrams per deciliter [mg/dL]) are presented categorical as follows:
  Protein: <10 (-)*; 10-25 (+-)*; 25-85 (+); 85-250 (2+); 250-800 (3+).
  Glucose: <30 (-)*; 30-60 (+-)*; 60-125 (+); 125-250 (2+); 250-750 (3+).
  Urobilinogen: <1.5 (+-)*; 1.5-3.5 (+); 3.5-7 (2+); 7-14 (3+).
  Bilirubin: <0.35 (-)*; 0.35-1.5 (+); 1.5-5 (2+); 5-12 (3+).
  Occult blood: <0.015 (-)*; 0.015-0.045 (+-); 0.045-015 (+); 0.15-0.75 (2+); >0.75 (3+).
  Ketone body: <2.5 (-)*; 2.5-7.5 (+-); 7.5-30 (+); 30-70 (2+); 70-125 (3+).
  Normal ranges indicated by asterix*.
Time Frame: At Month 0 and Month 7
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 519 | 521
Participants
  Protein (-) [Month 0] | 496 | 492
  Protein (+-) [Month 0] | 10 | 11
  Protein (+) [Month 0] | 9 | 16
  Protein (2+) [Month 0] | 2 | 1
  Protein (3+) [Month 0] | 1 | 1
  Protein (Unknown) [Month 0] | 1 | 0
  Protein (-) [Month 7] | 444 | 448
  Protein (+-) [Month 7] | 10 | 11
  Protein (+) [Month 7] | 11 | 14
  Protein (2+) [Month 7] | 1 | 1
  Protein (3+) [Month 7] | 0 | 0
  Protein (Unknown) [Month 7] | 53 | 47
  Glucose (-) [Month 0] | 513 | 520
  Glucose (+-) [Month 0] | 3 | 0
  Glucose (+) [Month 0] | 0 | 0
  Glucose (2+) [Month 0] | 0 | 1
  Glucose (3+) [Month 0] | 2 | 0
  Glucose (Unknown) [Month 0] | 1 | 0
  Glucose (-) [Month 7] | 459 | 471
  Glucose (+-) [Month 7] | 2 | 2
  Glucose (+) [Month 7] | 2 | 1
  Glucose (2+) [Month 7] | 3 | 0
  Glucose (3+) [Month 7] | 0 | 0
  Glucose (Unknown) [Month 7] | 53 | 47
  Urobilinogen (-) [Month 0] | 0 | 0
  Urobilinogen (+-) [Month 0] | 506 | 502
  Urobilinogen (+) [Month 0] | 11 | 15
  Urobilinogen (2+) [Month 0] | 1 | 2
  Urobilinogen (3+) [Month 0] | 0 | 2
  Urobilinogen (Unknown) [Month 0] | 1 | 0
  Urobilinogen (-) [Month 7] | 0 | 0
  Urobilinogen (+-) [Month 7] | 460 | 460
  Urobilinogen (+) [Month 7] | 6 | 12
  Urobilinogen (2+) [Month 7] | 0 | 1
  Urobilinogen (3+) [Month 7] | 0 | 1
  Urobilinogen (Unknown) [Month 7] | 53 | 47
  Occult Blood (-) [Month 0] | 483 | 495
  Occult Blood (+-) [Month 0] | 11 | 7
  Occult Blood (+) [Month 0] | 11 | 9
  Occult Blood (2+) [Month 0] | 9 | 8
  Occult Blood (3+) [Month 0] | 4 | 2
  Occult Blood (Unknown) [Month 0] | 1 | 0
  Occult Blood (-) [Month 7] | 393 | 398
  Occult Blood (+-) [Month 7] | 22 | 28
  Occult Blood (+) [Month 7] | 19 | 20
  Occult Blood (2+) [Month 7] | 22 | 18
  Occult Blood (3+) [Month 7] | 10 | 10
  Occult Blood (Unknown) [Month 7] | 53 | 47
  Ketone Body (-) [Month 0] | 501 | 506
  Ketone Body (+-) [Month 0] | 0 | 0
  Ketone Body (+) [Month 0] | 9 | 8
  Ketone Body (2+) [Month 0] | 7 | 6
  Ketone Body (3+) [Month 0] | 1 | 1
  Ketone Body (Unknown) [Month 0] | 1 | 0
  Ketone Body (-) [Month 7] | 452 | 460
  Ketone Body (+-) [Month 7] | 0 | 0
  Ketone Body (+) [Month 7] | 10 | 10
  Ketone Body (2+) [Month 7] | 3 | 3
  Ketone Body (3+) [Month 7] | 1 | 1
  Ketone Body (Unknown) [Month 7] | 53 | 47
  Bilirubin (-) [Month 0] | 517 | 520
  Bilirubin (+-) [Month 0] | 0 | 0
  Bilirubin (+) [Month 0] | 1 | 1
  Bilirubin (2+) [Month 0] | 0 | 0
  Bilirubin (3+) [Month 0] | 0 | 0
  Bilirubin (Unknown) [Month 0] | 1 | 0
  Bilirubin (-) [Month 7] | 466 | 474
  Bilirubin (+-) [Month 7] | 0 | 0
  Bilirubin (+) [Month 7] | 0 | 0
  Bilirubin (2+) [Month 7] | 0 | 0
  Bilirubin (3+) [Month 7] | 0 | 0
  Bilirubin (Unknown) [Month 7] | 53 | 47

ADVERSE EVENTS:
Time Frame: - For serious adverse events: thoughout the study period (up to Month 24). - For other adverse events: -- during the 30-day (non-systematically assessed) or -- during the 7-day (systematically assessed) follow-up period after any vaccination.
Description: Total number of subjects at risk corresponds to
  * all subjects in the Total Vaccinated Cohort for serious events and non-systematically assessed other events;
  * those subjects in the Total Vaccinated Cohort with at least one documented dose.
Arm/Group | Cervarix Group | Aimmugen Group
All-Cause Mortality (participants affected / at risk) | 1/519 | 0/521
Serious Adverse Events (participants affected / at risk) | 18/519 | 19/521
Other Adverse Events (participants affected / at risk) | 512/519 | 459/521
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=519) | Aimmugen Group (N=521)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 3
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Allergic granulomatous angiitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Mastitis postpartum (Infections and infestations) | 0 | 1
Moyamoya disease (Nervous system disorders) | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Group (N=519) | Aimmugen Group (N=521)
Pain (General disorders) | 508/512 | 214/510
Redness (General disorders) | 455/512 | 287/510
Swelling (General disorders) | 401/512 | 165/510
Arthralgia (General disorders) | 123/512 | 61/511
Fatigue (General disorders) | 341/512 | 300/511
Fever (General disorders) | 41/512 | 28/511
Gastrointestinal symptoms (General disorders) | 172/512 | 167/511
Headache (General disorders) | 250/512 | 222/511
Myalgia (General disorders) | 262/512 | 128/511
Rash (General disorders) | 33/512 | 24/511
Nasopharyngitis (Infections and infestations) | 110 | 91
Injection site pruritus (General disorders) | 83 | 15
Injection site warmth (General disorders) | 69 | 6
Headache (Nervous system disorders) | 19 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.